CLINICAL TRIAL: NCT03111732
Title: A Phase 2 Study of Pembrolizumab, a Monoclonal Antibody Against PD-1, in Combination With Capecitabine and Oxaliplatin (CAPOX) in Subjects With Advanced Biliary Tract Carcinoma (BTC)
Brief Title: Pembrolizumab, a Monoclonal Antibody Against PD-1, in Combination With Capecitabine and Oxaliplatin (CAPOX) in People With Advanced Biliary Tract Carcinoma (BTC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., National Cancer Institute, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170082; 17-C-0082
Record Dates: First submitted 2017-04-12; First posted 2017-04-13 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Biliary Tract Neoplasms; Cholangiocarcinoma; Bile Duct Cancer; Liver Cancer; Gallbladder Cancer
Keywords: Immune-Based Strategies; Anti-PD1 Therapy; Chronic Inflammation; Combination Chemotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms; Liver Neoplasms; Gallbladder Neoplasms | interventions — pembrolizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1/Arm 1 (Experimental): Pembrolizumab plus Oxaliplatin plus Capecitabine
  Interventions: Biological: Pembrolizumab (MK-3475); Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Biological: Pembrolizumab (MK-3475) — 200 mg will be administered as an IV infusion on Day 1 of each 21 day cycle
Drug: Oxaliplatin — 130mg/m(2) IV Infusion will be administered as an IV infusion on Day 1 of cycles 1-6
Drug: Capecitabine — 750 mg/m(2) will be administered orally twice a day on Days 1-14 of cycles 1-6

SUMMARY:
Background:

Biliary tract cancers are rare but they are serious. Researchers want to see if a certain drug helps the immune system fight cancer cells. The drug is called pembrolizumab. It may work even better with two chemotherapy drugs that are widely used to treat gastrointestinal cancers.

Objective:

To study if pembrolizumab given with capecitabine and oxaliplatin (CAPOX) increases the time it takes for a person's biliary tract cancer to get worse.

Eligibility:

People age 18 and older with previously treated biliary tract cancer that has spread to other parts of the body

Design:

Participants will be screened with tests as part of their regular cancer care.

Each study cycle is 3 weeks.

For 6 cycles, participants will:

Get pembrolizumab and oxaliplatin on day 1 of each cycle. They will be given in an intravenous (IV) catheter.

Take capecitabine by mouth for 2 weeks then have 1 week without it.

Participants will complete a patient diary.

Starting with cycle 7, participants will get only pembrolizumab. They will get it once every 3 weeks.

On day 1 of every cycle, participants will have:

Physical exam

Review of symptoms and how well they do normal activities

Blood tests

Every 9 weeks, they will have a scan.

Participants may have tumor samples taken.

Participants will have a final visit about 1 month after they stop the study drug. After that, they will be contacted by phone or email yearly.

DETAILED DESCRIPTION:
Background:

* The most compelling argument in favor of testing immune-based strategies (and anti-Programmed cell death protein 1 (PD1) therapy in particular) in biliary tract cancers (BTC) is that chronic inflammation appears to be the most common etiologic factor in the development of biliary tract cancer.
* Single-agent activity has been shown for PD1-directed therapy in BTC. Given the potential for oxaliplatin-induced immunogenic cell death we would like to evaluate the combination of capecitabine and oxaliplatin (CAPOX) chemotherapy with pembrolizumab.

Objective:

To determine the 5-month progression free survival (PFS) of Pembrolizumab in combination with CAPOX in patients with advanced biliary tract carcinoma.

Eligibility:

* Histologically confirmed diagnosis biliary tract carcinoma OR histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of biliary tract carcinoma.
* Patients must have at least one prior chemotherapeutic regimen.
* Patients must have disease that is not amenable to potentially curative resection.
* No prior treatment with oxaliplatin.

Design:

The proposed study is a phase II study of Pembrolizumab in combination with CAPOX in patients with advanced biliary tract carcinoma

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histopathological confirmation of biliary tract carcinoma (BTC) by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study OR histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of biliary tract carcinoma. The term BTC includes intra- or extrahepatic cholangiocarcinoma, gallbladder cancer or ampullary cancer.
* Patients must have disease that is not amenable to potentially curative resection. Patients must have received, been intolerant of or refused at least one line of chemotherapy.
* Patients must have at least one focus of measurable metastatic disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patients must have at least one focus of metastatic disease that is amenable to pre- and on-treatment biopsies. Ideally the biopsied lesion should not be one of the target measurable lesions, although this can be up to the discretion of the investigators.
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 2 xULN
  * Serum albumin greater than or equal to 2.5g/dl
  * Patients are eligible with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) up to 5 x upper limit of normal (ULN).
  * creatinine <1.5X institution upper limit of normal OR creatinine clearance greater than or equal to 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.
* Patients must not have other invasive malignancies within the past 5 years (with the exception of non-melanoma skin cancers, non-invasive bladder cancer or localized prostate cancer for whom systemic therapy is not required).
* Patient must be able to understand and willing to sign a written informed consent document.
* The effects of Pembrolizumab in combination with Capecitabine and Oxaliplatin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and up to 120 days after the last dose of the drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

* Patients who have had standard of care chemotherapy, large field radiotherapy, or major surgery must wait 2 weeks prior to entering the study.
* Previous treatment with immune checkpoint inhibitors.
* Patients who have undergone prior liver transplantation are ineligible.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations that would limit compliance with study requirements.
* History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* History of chronic autoimmune disease (e.g., Addison s disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, rheumatoid arthritis, hypophysitis, etc.) with symptomatic disease within the 3 years before randomization. Note: Active vitiligo or a history of vitiligo will not be a basis for exclusion.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of Information and Consent and compliance with the requirements of the protocol
* Active or history of inflammatory bowel disease (colitis, Crohn's), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegener's granulomatosis.
* Currently receiving immunosuppressive doses of steroids or other immunosuppressive medications (inhaled and topical steroids are permitted)
* History of sarcoidosis syndrome.
* Known history of active tuberculosis.
* Patients should not be vaccinated with live attenuated vaccines within 1 month of starting pembrolizumab treatment.
* Active hepatitis B or C infection.
* Human Immunodeficiency Virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and pembrolizumab. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that pembrolizumab may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events.
* History of hypersensitivity reaction to human or mouse antibody products.
* Female patients who are pregnant or breastfeeding. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Pembrolizumab in combination with Capecitabine and Oxaliplatin, breastfeeding should be discontinued.
* Patients with unhealed surgical wounds for more than 30 days.
* Prior therapy with oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2021-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Lamarca A, Hubner RA, David Ryder W, Valle JW. Second-line chemotherapy in advanced biliary cancer: a systematic review. Ann Oncol. 2014 Dec;25(12):2328-2338. doi: 10.1093/annonc/mdu162. Epub 2014 Apr 25. PMID 24769639
- [Derived] Monge C, Pehrsson EC, Xie C, Duffy AG, Mabry D, Wood BJ, Kleiner DE, Steinberg SM, Figg WD, Redd B, Budhu A, Wang S, Tandon M, Ma L, Wei Wang X, Greten TF. A Phase II Study of Pembrolizumab in Combination with Capecitabine and Oxaliplatin with Molecular Profiling in Patients with Advanced Biliary Tract Carcinoma. Oncologist. 2022 Mar 11;27(3):e273-e285. doi: 10.1093/oncolo/oyab073. PMID 35274717
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0082.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine: Pembrolizumab plus Oxaliplatin plus Capecitabine
  Pembrolizumab (MK-3475): 200 mg will be administered as an intravenous (IV) infusion on Day 1 of each 21 day cycle
  Oxaliplatin: 130mg/m(2) IV Infusion will be administered as an IV infusion on Day 1 of cycles 1-6
  Capecitabine: 750 mg/m(2) will be administered orally twice a day on Days 1-14 of cycles 1-6
Period: Overall Study
Arm/Group | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine
Started | 11
Completed | 6
Not Completed | 5
Not completed — Enrolled in different study | 1
Not completed — Progressive disease | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.32 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Median amount of time subject survives without disease progression for 5 months after treatment. Disease progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: 5 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine
Number analyzed (Participants) | 11
Months | 4.54 [2.5 to 9.6]

2. Secondary Outcome: Number of Participants Obtaining a Complete Response (CR) and Partial Response (PR)
Description: Number of participants obtaining CR and PR per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria of all evaluable patients. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions,taking as reference the baseline sum of diameters.
Time Frame: Every 9 Weeks, until disease progression or patient is taken off the trial, whichever comes first, approximately 36 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine
Number analyzed (Participants) | 11
Participants
  Complete Response | 0
  Partial Response | 3

3. Secondary Outcome: Overall Survival
Description: Median amount of time subject survives after therapy.
Time Frame: Death, approximately 48 weeks after stopping therapy.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine
Number analyzed (Participants) | 11
Weeks | 43 [22 to 66]

4. Secondary Outcome: Number Participants With Grade 1-4 Adverse Events Unrelated, Unlikely, Possibly, Probably and Definitely Related to Pembrolizumab
Description: Here is the number of participants with grade 1-4 adverse events unrelated, unlikely, possibly, probably and definitely related to study drug assessed by the Common Terminology Criteria for Adverse Events v4.0. Mild (Grade1), moderate (Grade 2), severe (Grade 3), and life-threatening or disabling (Grade 4).
Time Frame: 30 Days After Enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Unrelated: Unrelated to drug.
- Unlikely: Unlikely related to drug.
- Possibly: Possibly related to drug.
- Probably: Probably related to drug.
- Definitely: Definitely related to drug.
Arm/Group | Unrelated | Unlikely | Possibly | Probably | Definitely
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
Participants
  Grade 1 | 9 | 11 | 10 | 3 | 0
  Grade 2 | 7 | 10 | 8 | 3 | 0
  Grade 3 | 3 | 7 | 8 | 1 | 0
  Grade 4 | 0 | 3 | 2 | 0 | 0

5. Secondary Outcome: Number Participants With Grade 1-4 Adverse Events Unrelated, Unlikely, Possibly, Probably and Definitely Related to Oxaliplatin
Description: as for outcome 4
Time Frame: 30 Days After Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated | Unlikely | Possibly | Probably | Definitely
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
Participants
  Grade 1 | 9 | 11 | 11 | 7 | 4
  Grade 2 | 6 | 10 | 9 | 5 | 2
  Grade 3 | 3 | 6 | 8 | 2 | 0
  Grade 4 | 0 | 2 | 2 | 1 | 0

6. Secondary Outcome: Number of Participants With Grade 1-4 Adverse Events Unrelated, Unlikely, Possibly, and Probably Related to Capecitabine
Description: Here is the number of participants with grade 1-4 adverse events unrelated, unlikely, possibly, and probably related to study drug assessed by the Common Terminology Criteria for Adverse Events v4.0. Mild (Grade1), moderate (Grade 2), severe (Grade 3), and life-threatening or disabling (Grade 4).
Time Frame: 30 Days After Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated | Unlikely | Possibly | Probably | Definitely
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
Participants
  Grade 1 | 9 | 11 | 11 | 6 | 0
  Grade 2 | 7 | 9 | 9 | 4 | 0
  Grade 3 | 3 | 6 | 7 | 2 | 0
  Grade 4 | 0 | 2 | 2 | 1 | 0

7. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 38 months and 25 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 38 months and 25 days.
Arm/Group | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine
All-Cause Mortality (participants affected / at risk) | 9/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine (N=11)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Infections and infestations - Other, unknown origin (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm 1 - Pembrolizumab Plus Oxaliplatin Plus Capecitabine (N=11)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (8)
Activated partial thromboplastin time prolonged (Investigations) | 5 (6)
Alanine aminotransferase increased (Investigations) | 9 (13)
Alkaline phosphatase increased (Investigations) | 7 (12)
Anemia (Blood and lymphatic system disorders) | 8 (25)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 9 (18)
Autoimmune disorder (Immune system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (2)
Blood bilirubin increased (Investigations) | 6 (12)
Blurred vision (Eye disorders) | 1 (1)
Chills (General disorders) | 5 (5)
Colitis (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Creatinine increased (Investigations) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (17)
Dizziness (Nervous system disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dysesthesia (Nervous system disorders) | 6 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye disorders - Other, Conjunctival hemorrhage (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 6 (10)
Fever (General disorders) | 5 (9)
Flu like symptoms (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Cramping (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, indigestion (Gastrointestinal disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 5 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (12)
Immune system disorders - Other, Adrenal insufficiency (Immune system disorders) | 1 (1)
Infections and infestations - Other, Herpes labialis (Infections and infestations) | 1 (1)
Infections and infestations - Other, Mucositis (Infections and infestations) | 1 (1)
Infections and infestations - Other, Thrush - tongue, mucosal infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, Erythema, swelling under bilat. Eyes (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lipase increased (Investigations) | 1 (6)
Lymphocyte count decreased (Investigations) | 11 (51)
Malaise (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6)
Neutrophil count decreased (Investigations) | 5 (13)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 4 (7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (17)
Platelet count decreased (Investigations) | 9 (20)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Serum amylase increased (Investigations) | 5 (13)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Thrush- mouth (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Erythema, swelling under bilat. Eyes (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Rash, nose (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Skin lesion- cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Swelling- lower leg (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, brittle nails (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, buttocks (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, swelling - left foot (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 8 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT03111732/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT03111732/ICF_001.pdf